CLINICAL TRIAL: NCT05324644
Title: The Effect of Motivational Interview Attempt on Self-Efficacy Level and Decision to Quit Smoking of University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Green Crescent (Yeşilay) (Unknown)
Responsible Party: Principal Investigator, Feyza Dereli, Lecturer, Izmir Katip Celebi University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1071
Record Dates: First submitted 2022-04-06; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Codependency, Psychological
Keywords: motivational interview, quit smoking, behavior change
MeSH Terms: conditions — Codependency, Psychological | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: This study is a randomized and case-control study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): 32 randomly selected first-year students in the university, who voluntarily agreed to be recruited into the study and smoke and are considering quitting.
  Interventions: Behavioral: Motivational interview
- Control group (No Intervention): 32 randomly selected first-year students in the university, who voluntarily agreed to be recruited into the study and smoke and are considering quitting.

INTERVENTIONS:
Behavioral: Motivational interview — In the first interviews with the students; It is planned to provide information about acquaintance and research, fill in the scales in 10-15 minutes, make CO measurements, and also conduct an average of 20-40 minutes of motivational interviews in the intervention group. In the second interview in the 1st month, it is planned to summarize the first interview, fill in the scales in 3-5 minutes, make the CO measurements in 10-15 minutes or get the measurement results and apply motivational interview in the average of 20-40 minutes. In the third interview in the 3rd month, it is planned to summarize the second interview in 3-5 min, fill in the scales in 10-15 minutes, make CO measurements or get the measurement results and to apply motivational interviews for an average of 20-40 minutes. In the last interview in the 6th month, it is planned to summarize the 3rd-month interview, to apply the scales for approximately 10-15 minutes, to make CO measurements or to get the measurement results.
  Arms: Interventional group

SUMMARY:
This study aimed to determine the effect of motivational interview initiatives on the smoking cessation decisions of university students. In this study, which will be conducted as a randomized, case-control study; Student introduction form, Fagerström Nicotine Addiction Test, Decision-Making Balance Scale, Self-efficacy adequacy scale, Behavior Change Stage Diagnosis Short Questionnaire, Beck Depression Scale, Smoking Desire Scale will be used, CO will be measured. Motivational interview initiative will be applied to first-year students who are enrolled in the university, who smoke and are considering quitting. The estimated duration of the study is 8-10 months. Maximum number of volunteers will be 60.

DETAILED DESCRIPTION:
More than 7 million people in the world and more than 100,000 people in Turkey die from diseases related to tobacco use annually. Young people are one of the most important target groups of the tobacco industry. For these reasons, one of the goals in the international and national (Tobacco Control Strategy Document and Action Plan 2018-2023 for Turkey) tobacco control programs is to include protective, preventive and therapeutic studies, especially for children and youth. Currently, there are two treatment approaches recommended for smoking cessation. They are pharmacological treatment and behavioural treatment/motivation. The aim of this study is to evaluate the effect of the motivational interview initiative on the self-efficacy level of university students and their decision to quit smoking.

The research will be conducted in a randomized, intervention-control group experimental research design. The study will be carried out on first-year students of a university. The universe of the research; 1st-year students (N: 4543) registered in the 2020-2021 academic year. The number of students to be reached after the announcement was determined as 358 by using the 72% value, which is the result of the smoking status determination survey conducted at the same university in the 2019-2020 academic year in the previous year, using the sample calculation method with the known universe.

The study will be announced on the website of the university where the research will be conducted for first-year students who smoke and want to quit. Students who want to participate, who have not been diagnosed with depression and whose Beck depression score is mild and minimally depressed will constitute the sample group.

The sample size was calculated using power analysis. Self-efficacy and efficacy score effect size between intervention and control was calculated as 0.49 and n=23 students from each group were calculated, with a 0.05 margin of error and Power of 83.83%. As a result of the sample number calculation, 23 intervention and 23 control group students should be included. Considering that there may be losses in the later stages of the study, 40 students will be included in the study for each group. In line with the feasibility of education and training during the pandemic process, face-to-face and online interviews will be held with the hybrid interview method. Students willing to quit smoking will be divided into control and intervention groups using the simple random sampling technique according to the random numbers assignment list created in the Excel program by the biostatistics expert. In order to avoid bias, students will not be informed about which group they are in by using the single-blind study technique.

Motivational interviews and related scales will be applied to the students in the initiative group and CO measurement will be made. In cases where it is not appropriate to measure CO due to pandemic conditions, students will not be able to measure it. Such cases will be recorded in the data collection form.

After the research, motivational interviews will be made to the students in the control group who want to support their decision to quit smoking.

The researcher who will conduct the interviews has received motivational interview technique training. For the individual motivational interview to be held with the students in the intervention group, the researcher will make the first interview by determining the appropriate times with the students. Afterwards, motivational interviews will be held at the 1st, 3rd and 6th months, in which relapses and behavioural changes are evaluated (Behavioral Change Stage Diagnosis Short Questionnaire). Interviews are planned to be conducted using a hybrid method (face-to-face or online).

In the first of the individual interviews with the students; It is planned to provide information about acquaintance and research, fill in the scales in 10-15 minutes, make and evaluate CO measurements, and also conduct an average of 20-40 minutes of motivational interviews in the intervention group. In the second interview in the 1st month, it is planned to summarize the first interview, fill in the scales in 3-5 minutes, make the CO measurements in 10-15 minutes or get the measurement results and apply a motivational interview in the average of 20-40 minutes. In the third interview in the 3rd month, it is planned to summarize the second interview in 3-5 min, fill in the scales in 10-15 minutes, make CO measurements or take the measurement results made by the students in the smoking cessation polyclinics and to apply motivational interviews for an average of 20-40 minutes. In the last interview in the 6th month, it is planned to summarize the 3rd-month interview, to apply the scales to both groups for approximately 10-15 minutes, to make CO measurements or to get the measurement results.

ELIGIBILITY:
Inclusion Criteria:

1. Students in Year 1
2. Smoker,
3. 18 years and older,
4. Those who have not received a psychiatric diagnosis made by the physician,
5. Those who want to quit smoking,
6. Volunteer students who accept the motivational interview.

Exclusion Criteria:

1. Non-smokers,
2. 18 years old and under,
3. Taking the course of the researcher teacher due to vulnerability,
4. Students who do not want to participate voluntarily will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of people who quit smoking | Six months
  The number of people who quit smoking in the groups at the end of the study.

OTHER OUTCOMES:
Fagerström Test for Nicotine Dependence | Six months
  Fagerström Test for Nicotine Dependence
Decision Making Balance Scale | Six months
  Decision Making Balance Scale
Self-efficacy adequacy scale | Six months
  Self-efficacy adequacy scale
Behavior Change Stage Diagnosis Short Questionnaire | Six months
  Behavior Change Stage Diagnosis Short Questionnaire
Smoking desire scale | Six months
  Smoking desire scale
CO Measurement | Six months
  CO Measurement

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akdur, R. Gençlerde Sigara Salgını (2010). Ankara Üniversitesi Tıp Fakültesi Halk Sağlığı Yayınları. Ankara
- [Background] Apodaca TR, Abrantes AM, Strong DR, Ramsey SE, Brown RA. Readiness to change smoking behavior in adolescents with psychiatric disorders. Addict Behav. 2007 Jun;32(6):1119-30. doi: 10.1016/j.addbeh.2006.07.016. Epub 2006 Sep 1. PMID 16950572
- [Background] Demirezen M, Kurcer MA. Questionnaire of smoking urges Turkish validity and reliability. TAF Prev Med Bull 2016;15:1-4.
- [Background] DiClemente CC, Prochaska JO, Fairhurst SK, Velicer WF, Velasquez MM, Rossi JS. The process of smoking cessation: an analysis of precontemplation, contemplation, and preparation stages of change. J Consult Clin Psychol. 1991 Apr;59(2):295-304. doi: 10.1037//0022-006x.59.2.295. PMID 2030191
- [Background] Doğan, DG,. Ulukol, B. (2010). Ergenlerin sigara içmesini etkileyen faktörler ve sigara karşıtı iki eğitim modelinin etkinliği. İnönü Üniversitesi Tıp Fakültesi Dergisi.79-85.
- [Background] Edwards, L.K. (1993). Applied Analysis of Variance in the Behavior Sciences. Marcel Dekker. New York.
- [Background] 2008 PHS Guideline Update Panel, Liaisons, and Staff. Treating tobacco use and dependence: 2008 update U.S. Public Health Service Clinical Practice Guideline executive summary. Respir Care. 2008 Sep;53(9):1217-22. No abstract available. PMID 18807274
- [Background] Folkman S, Lazarus RS. An analysis of coping in a middle-aged community sample. J Health Soc Behav. 1980 Sep;21(3):219-39. No abstract available. PMID 7410799
- [Background] Gözüm S, Aksayan S. (1999). Öz-etkililik-yeterlik ölçeği'nin türkçe formunun güvenilirlik ve geçerliliği. Journal of Anatolia Nursing and Health Sciences;2(1):21-34.
- [Background] Health New Zeland. (2009). Testing for Carbon Monoxide in exhaled breath. (2020). Erişim adresi: http://www.healthnz.co.nz/CObreath.htm.
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Hisli, N. (1989). Beck depresyon envanterinin üniversite öğrencileri için geçerliği, güvenirliği. Psikoloji Dergisi, 7(23), 3-13.
- [Background] Kamışlı Özcan, S. (2007). Psikoeğitimsel Bir Programla Hemşirelerin Sigara Bırakma Durumları. Hacettepe Üniversitesi Sağlık Bilimleri Enstitüsü, Doktora Tezi. Ankara.
- [Background] Karadağlı, F., Nahcivan, N. (2012). Sigara içen bireylerde sigara bırakmaya hazıroluşluk durumu ile ilişkili faktörler. DEUHYO Dergisi, 5(1), (s. 8- 15).
- [Background] Karagöz Y. SPSS 21.1 (2014). Uygulamalı Biyoistatistik. İstanbul: Nobel Tıp Kitabevi; .s.1-740.
- [Background] Kaya N, Çilli AS. (2002). Üniversite Öğrencilerinde Nikotin, Alkol ve Madde Bağımlılığının On iki Aylık Yaygınlığı, Bağımlılık Dergisi 3(2).
- [Background] Kisioğlu N, Öztürk M, Doğan M. (2002). Süleyman Demirel Üniversitesi İlk ve Son Sınıf Öğrencilerinin Sigaraya Yönelik Bilgi, Tutum, Davranışları ve Sigaraya Başlama ve Alışma Durumları.
- [Background] Lancaster T, Stead L, Silagy C, Sowden A. Effectiveness of interventions to help people stop smoking: findings from the Cochrane Library. BMJ. 2000 Aug 5;321(7257):355-8. doi: 10.1136/bmj.321.7257.355. No abstract available. PMID 10926597
- [Background] Mueller, K. E., and Barton, C. N. (1989). 'Approximate Power for Repeated-Measures ANOVA Lacking Sphericity. Journal of the American Statistical Association, Volume 84, No. 406, pages 549-555.
- [Background] Muller KE, Lavange LM, Ramey SL, Ramey CT. Power Calculations for General Linear Multivariate Models Including Repeated Measures Applications. J Am Stat Assoc. 1992 Dec 1;87(420):1209-1226. doi: 10.1080/01621459.1992.10476281. PMID 24790282
- [Background] Ögel K. (2009). Motivasyonel görüşme tekniği. Türkiye Klinikleri Journal of Psychiatry-Special Topics 2009;2(2):41-44.
- [Background] Onur ST, Uysal MA, Iliaz S, Yurt S, Bahadir A, Hattatoglu DG, Ortakoylu MG, Bagci BA, Chousein EG. Does Short Message Service Increase Adherence to Smoking Cessation Clinic Appointments and Quitting Smoking? Balkan Med J. 2016 Sep;33(5):525-531. doi: 10.5152/balkanmedj.2016.151610. Epub 2016 Sep 1. PMID 27761280
- [Background] Özdemir H, Taşcı S. (2013). Motivasyonel görüşme tekniği ve hemşirelikte kullanımı. ERÜ Sağlık Bilimleri Fakültesi Dergisi;1(1):41-47.
- [Background] Pardavila-Belio MI, Garcia-Vivar C, Pimenta AM, Canga-Armayor A, Pueyo-Garrigues S, Canga-Armayor N. Intervention study for smoking cessation in Spanish college students: pragmatic randomized controlled trial. Addiction. 2015 Oct;110(10):1676-83. doi: 10.1111/add.13009. Epub 2015 Jul 2. PMID 26053958
- [Background] Prochazka AV. New developments in smoking cessation. Chest. 2000 Apr;117(4 Suppl 1):169S-175S. doi: 10.1378/chest.117.4_suppl_1.169s. PMID 10777474
- [Background] Uysal MA, Kadakal F, Karsidag C, Bayram NG, Uysal O, Yilmaz V. Fagerstrom test for nicotine dependence: reliability in a Turkish sample and factor analysis. Tuberk Toraks. 2004;52(2):115-21. PMID 15241694
- [Background] Yalcinkaya-Alkar O, Karanci AN. What are the differences in decisional balance and self-efficacy between Turkish smokers in different stages of change? Addict Behav. 2007 Apr;32(4):836-49. doi: 10.1016/j.addbeh.2006.06.023. Epub 2006 Jul 13. PMID 16842929
- See also: Green crescent — https://www.yesilay.org.tr/tr